CLINICAL TRIAL: NCT03051529
Title: Combined Spinal- Epidural Anesthesia (CSE) for Vascular and Orthopedic Operations in Patients With Dilated Cardiomyopathy
Brief Title: Combined Spinal- Epidural Anesthesia in Patients With Dilated Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Other Study IDs: IRB00009900
Record Dates: First submitted 2016-03-16; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- combined spinal epidural: 24 patients with dilated cardiomyopathy undergoing vascular surgery in the lower half of the body under combined spinal epidural anesthesia will be enrolled in the study
  Interventions: Other: combined spinal epidural anesthesia

INTERVENTIONS:
Other: combined spinal epidural anesthesia — After approval by local research ethics committee of the Faculty of Medicine, and informed written consent obtained from all patients, 24 patients having dilated cardiomyopathy, subjected to vascular surgery in the lower half of the body under CSEA

SUMMARY:
This study was conducted on 24 patients who have ischemic dilated cardiomyopathy, underwent non cardiac surgery in the lower half of the body under the effect of combined spinal epidural anesthesia at Assiut university hospital. Intraoperative Hemodynamic monitoring including invasive blood pressure, heart rate, and CVP was established, in addition to pre and postoperative, 12 lead ECG, echocardiography, and venous sampling for Brain natriuretic peptide measurement were done .

This study tried to assess the safety of this anesthetic technique on such group of cardiac patients along over the hospital stay period and up to 6 months postoperatively, in addition to the predictability of Brain natriuretic peptide as a cardiac biomarker regarding to the major adverse cardiac events and cardiac mortality for these group of patients .

DETAILED DESCRIPTION:
Dilated cardiomyopathy (DCM) is characterized by ventricular dilatation and impaired systolic cardiac function. Anesthetic management, of patients with cardiomyopathy with reduced systolic function, is challenging and may be associated with high mortality.

Objective: The purpose of this study was to evaluate the hemodynamic effects of combined spinal epidural anesthesia (CSEA) in patients with dilated cardiomyopathy, underwent vascular surgery in the lower half of the body, in addition to assess the safety of this anesthetic technique in the early postoperative period.

Method: After approval by local research ethics committee of the Faculty of Medicine, and informed written consent obtained from all patients, 24 patients having dilated cardiomyopathy, subjected to vascular surgery in the lower half of the body under CSEA. The effects of CSEA on hemodynamics; IBP, HR and CVP (measured at base line and then every 10 min), in addition to cardiac complications during the hospital stay period were studied.

ELIGIBILITY:
Inclusion Criteria:

* 24 patients Cardiomyopathy DCM underwent infra-inguinal vascular surgery under the effect of combined spinal epidural technique were included in a prospective trial single center observational study.

Exclusion Criteria:

* Patients with significant fluid and electrolyte imbalance, major arrhythmias or heart failure or unstable angina, systolic blood pressure at rest < 100 mmHg, heart rate < 50, serum creatinine >2.0 mg /dl, and patients who required emergency surgery were excluded from the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 patients having dilated cardiomyopathy, subjected to vascular surgery in the lower half of the body under combined spinal epidural anesthesia CSEA.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
early postoperative cardiac complications | 7 days post operative
  following up the patients for cardiac events such as arrhythmia , heart failure , new ischemic cardiac events

SECONDARY OUTCOMES:
BNP level changes | 72 hours postoperative
  BNP follow up

IPD SHARING:
Plan to Share IPD: No